CLINICAL TRIAL: NCT02966119
Title: Evaluation of the Benefit/Risk Ratio of Restarting or Avoiding Antiplatelet Drugs in Patients Who Had a Spontaneous Intracerebral Hemorrhage While Treated With Antithrombotic Drugs : RESTART-FR Study
Brief Title: REstart or STop Antithrombotic Randomised Trial in France
Acronym: RESTART-Fr
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Lille (Other)
Collaborators: Région Hauts de France, France (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015_11; 2015-A01319-40 (Other: ID-RCB number, ANSM); PHRCI_2014 (Other: PHRC number, DGOS)
Record Dates: First submitted 2016-07-13; First posted 2016-11-17 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Hemorrhage
Keywords: stroke; intracranial hemorrhage; intracerebral hemorrhage; antithrombotic drugs; brain microbleeds
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Intracranial Hemorrhages | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Start antiplatelet drug(s) (Experimental): If the patient is randomized in this arm, an antiplatelet agent (aspirin or clopidogrel or dypyridamole), chosen by the patient's physician before the randomisation, will be prescribed to the patient during the study period
  Interventions: Drug: Clopidogrel or Aspirin and/or Dypyridamole
- Avoid antiplatelet drug(s) (No Intervention): If the patient is randomized in this arm, antiplatelet drugs will not be prescribed to the patient during the entire study period

INTERVENTIONS:
Drug: Clopidogrel or Aspirin and/or Dypyridamole — The physician will prescribe on this antiplatelet agent if the patient is randomized in the arm " restart"
  Arms: Start antiplatelet drug(s)

SUMMARY:
RESTART- fr is a randomised controlled trial for adults surviving spontaneous intracerebral haemorrhage who had taken an antithrombotic drug (i.e. anticoagulant or antiplatelet medication) for the prevention of vaso-occlusive disease before the ICH.

RESTART- fr is testing whether a policy of starting antiplatelet drugs (one or more of aspirin, clopidogrel, or dipyridamole, chosen at investigator's discretion) results in a beneficial net reduction of all serious vascular events over two years compared with a policy of avoiding antiplatelet drugs.

DETAILED DESCRIPTION:
More than one third of the adults with a stroke due to bleeding into the brain - known as brain haemorrhage - are taking drugs to prevent clotting when they have a brain haemorrhage.

These patients had previously suffered illnesses like angina, heart attack, or stroke due to blood vessel blockage, which is why they are treated with drugs to prevent further clots occurring. These drugs are usually stopped when the brain haemorrhage occurs.

But when patients recover from brain haemorrhage, they and their doctors are often uncertain about whether to restart these drugs to prevent further clots occurring, or whether to avoid them in case they increase the risk of brain haemorrhage happening again.

In this preliminary study of 292 such people who survive a brain haemorrhage, we will study the potentially beneficial effects of three antiplatelet drugs (one or more of aspirin, clopidogrel, or dipyridamole, chosen by the patient's physician) on the risks of heart attack, stroke and other clotting problems as well as their effect on the risk of a brain haemorrhage happening again.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 years.
* Spontaneous intracerebral hemorrhage confirmed by imaging
* Patient had been taken antithrombotic drug(s) for the prevention of vaso-occlusive disease for at least 1 week before ICH onset
* Randomisation more than 24 hours after ICH onset.
* Patient and their doctor are uncertain about whether to start or avoid antiplatelet drugs.
* Brain imaging that first diagnosed the ICH is available. Participant or representative consent.

Exclusion Criteria:

* intracerebral hemorrhage associated with : a vascular malformation (AVM, arterial aneurysm, cavernoma); a secondary hemorrhagic infarction; a cerebral venous thrombosis; a tumor
* Patients with a formal indication of restarting oral anticoagulants despite the ICH (eg mechanical heart valves or pulmonary embolism under 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with symptomatic intracerebral hemorrhage | at one year
  Occurrence of a fatal or non-fatal symptomatic ICH proven radiologically at follow-up ( brain CT or MRI) .

SECONDARY OUTCOMES:
serious fatal vascular events (i.e. followed by death within 30 days ) or non- fatal | at one year and at the end of follow-up (2 years)
  symptomatic hemorrhagic events, symptomatic ischemic events, stroke of undetermined nature
Other fatal events | at one year and at the end of follow-up (2 years)
  Death without pre-defined vascular cause
Rankin Scale | 2 years
  modified Rankin Scale: dichotomized mRS 0-1-2 (no dependency) versus 3 or more (dependency or death)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte CORDONNIER, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Yes
we plan to make IPD analysis with sister trial: RESTART UK

REFERENCES:
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Cheng X, Dong Q. Towards individualised secondary prevention after intracerebral haemorrhage. Lancet Neurol. 2021 Jun;20(6):411-413. doi: 10.1016/S1474-4422(21)00130-7. No abstract available. PMID 34022160